CLINICAL TRIAL: NCT01805011
Title: Study on Normal Ranges of Lipids in Breast Milk of Healthy Mothers
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 11.08.INF
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Mothers
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 50 healthy mothers
  Interventions: Other: minimum 4 months of breastfeeding

INTERVENTIONS:
Other: minimum 4 months of breastfeeding

SUMMARY:
This trial is undertaken to better understand the ranges of functional components normally found in human milk. This will strengthen the scientific knowledge on breast-milk composition as a "gold standard".

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 37 and not above 42 weeks
* 18 years old ≤ Mother ≤ 40 years old
* 18.5 ≤ pre-pregnancy BMI ≤ 29
* Mothers willing to breastfeed for the first 4 months

Exclusion Criteria:

* Gestational diabetes
* HTA < 140/90
* Mothers who are smokers while breast-feeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy mothers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
levels of lipids | After 1 month of Breastfeeding
  The primary objective of this trial is to determine the levels of lipids normally found in the breast-milk of healthy lactating mothers

SECONDARY OUTCOMES:
profile and quantity of sugars | After 1 month of breastfeeding
  Secondary objectives include the measure of the profile and quantity of sugars found in human milk

CONTACTS AND LOCATIONS:
Overall Officials: Le Ye Lee, Assistant Professor, Principal Investigator — NUHS

REFERENCES:
- [Derived] Sprenger N, Lee LY, De Castro CA, Steenhout P, Thakkar SK. Longitudinal change of selected human milk oligosaccharides and association to infants' growth, an observatory, single center, longitudinal cohort study. PLoS One. 2017 Feb 9;12(2):e0171814. doi: 10.1371/journal.pone.0171814. eCollection 2017. PMID 28182762